CLINICAL TRIAL: NCT06697418
Title: The Effect of Physical Activity Level Evaluated by Wrist-wearable Devices on Cardiovascular Disease Risk and Other Outcomes in Peritoneal Dialysis Patients
Status: Enrolling by invitation | Type: Observational
Sponsor: Ruijin Hospital (Other)
Responsible Party: Principal Investigator, Xie Jingyuan, MD, chief physician, Ruijin Hospital
Other Study IDs: PACOPD
Record Dates: First submitted 2024-10-15; First posted 2024-11-20 (Actual); Last update posted 2024-11-20 (Actual); Status verified 2024-11

CONDITIONS: Peritoneal Dialysis; Cardiovascular Diseases; Myocardial Infarct; Heart Failure; Cognitive Disorders
Keywords: peritoneal dialysis; physical activities; wristband; cardiovascular risk; cognition
MeSH Terms: conditions — Cardiovascular Diseases; Myocardial Infarction; Heart Failure; Cognitive Dysfunction; Motor Activity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Active Group: The average daily physical activity measured by the fitness tracker is above 5,000 steps.
- Sedentary Group: The average daily physical activity measured by the fitness tracker is below 5,000 steps.

SUMMARY:
This study aims to explore how daily physical activity (PA) levels affect the heart health and cognitive function of patients on peritoneal dialysis (PD). Using a fitness tracker, the investigators will measure how much patients move during the day and see if lower activity levels are linked to a higher risk of heart disease or memory issues.

The study has two parts:

Part A: The investigators will evaluate 266 patients to understand their current PA levels and how these relate to heart health and cognitive function.

Part B: The investigators will follow the same patients over a year, measuring their activity at the beginning and after 12 months. The investigators will divide them into two groups-those who increase their PA and those whose PA decreases-and follow their heart health and memory function over two years.

The goal is to understand whether higher PA levels can reduce the risk of heart problems and memory issues in PD patients.

DETAILED DESCRIPTION:
Cardiovascular disease (CVD) is the leading cause of death in patients with chronic kidney disease (CKD), and cognitive impairment is also common in CKD patients. Previous studies have suggested an association between physical activity (PA) levels, CVD, and mild cognitive impairment. However, no relevant studies have been conducted in peritoneal dialysis (PD) patients, who are at high risk for both CVD and cognitive impairment. This study aims to measure the daily PA levels of PD patients using a wristband and analyze its impact on CVD and cognitive function in these patients.

The study consists of two parts:

Part A: A cross-sectional study, planning to enroll 266 patients. Demographic and baseline clinical data will be recorded, and PA will be assessed using the wrist-wearable devices. CVD will be evaluated using cardiac enzyme levels, N-terminal pro-B-type natriuretic peptide (NTpro-BNP), and echocardiography (UCG) parameters, while cognitive function will be assessed with the MMSE, MOCA and other scales. A multivariate logistic regression model will be used to analyze the correlation between PA and the prevalence of CVD and cognitive impairment.

Part B: A prospective cohort study. The enrolled patients will undergo repeated PA assessments using the wristband at months 0 and 12. Based on changes in PA from baseline, patients will be divided into an increased PA group and a decreased PA group. Both groups will be followed up to record major cardiovascular events and assess changes in left ventricular function and structure using cardiac enzyme levels, NTpro-BNP, and UCG indicators. Cognitive function will be evaluated using the MMSE, MOCA and other scales at months 0, 12, and 24 to assess changes in cognitive levels.

Expected Results: PA levels are expected to be associated with CVD and cognitive impairment in PD patients, with lower PA levels or decreased PA predicting a higher risk of new-onset CVD and cognitive impairment.

Primary Hypothesis: Lower PA levels are associated with increased CVD risk in PD patients, while higher PA levels or improvements in PA are associated with a lower risk of new-onset CVD.

Secondary Hypothesis: Lower PA levels are associated with increased cognitive impairment in PD patients, while higher PA levels or improvements in PA are associated with a lower risk of new-onset cognitive impairment.

ELIGIBILITY:
Inclusion Criteria:

1. 18 years old or above, under 75 years old
2. Receiving peritoneal dialysis treatment in Ruijin hospital for more than three months
3. Having the ability to walk independently
4. Willing to accept relevant training and sign informed consent

Exclusion Criteria:

1. Unable or unwilling to provide written informed consent;
2. Unwilling to cooperate with regular follow-up or telephone follow-up;
3. Evidence of liver damage (ALT, AST≥ 2 times the upper limit of normal);
4. Patients with newly diagnosed malignant tumors in the past year or undergoing radiotherapy or chemotherapy;
5. NYHA class III or IV congestive heart failure, myocardial infarction, stable or unstable angina;
6. New-onset stroke (within the past 3 months, including cerebral hemorrhage and cerebral infarction);
7. Severe mental illness or a diagnosis of dementia.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Receiving peritoneal dialysis treatment in Ruijin hospital for more than three months
Sampling Method: Non-Probability Sample
Enrollment: 266 (Estimated)
Dates: Start 2024-10-01 (Actual); Primary Completion 2024-10-01 (Actual); Study Completion 2026-10-31 (Estimated)

PRIMARY OUTCOMES:
Number of participants with Composite Endpoints of Cardiovascular Events | through study completion, an average of 3 months
  The composite endpoint of cardiovascular events includes cardiovascular death, non-fatal myocardial infarction, heart failure, stroke, valve replacement surgery, and coronary artery bypass surgery. Planning to establish a terminal endpoint assessment group to review the medical records of each patient, with two physicians independently assessing the endpoints for each case.

SECONDARY OUTCOMES:
Change from baseline in levels of high-sensitivity cardiac troponin I in 2 years | Baseline and the 12th, 24th month after entering the cohort
  Cardiac Troponin I (cTnI) is a highly specific biomarker used to assess myocardial injury. It is a subunit of the troponin complex that regulates cardiac muscle contraction. cTnI is uniquely expressed in cardiac muscle and is released into the bloodstream during myocardial cell damage, making it a critical indicator of myocardial injury. Levels of high-sensitivity cardiac troponin I will be evaluated in ug/L.
Change from baseline in levels of myoglobin in 2 years | Baseline and the 12th, 24th month after entering the cohort
  A heme-containing protein found in cardiac and skeletal muscle, released very early during muscle injury. Levels of myoglobin will be evaluated in ug/L.
Change from baseline in levels of Creatine Kinase-MB (CK-MB) in 2 years | Baseline and the 12th, 24th month after entering the cohort
  A cardiac-specific isoenzyme of CK, more specific to myocardial tissue than total CK. Levels of CK-MB will be evaluated in ug/L.
Change from baseline in levels of Creatine Kinase (CK) in 2 years | Baseline and the 12th, 24th month after entering the cohort
  An enzyme found in various tissues, including skeletal and cardiac muscles. It catalyzes ATP production during muscle contraction. Levels of CK will be evaluated in ug/L.
Change from baseline in levels of parameters from echocardiogram in 2 years | Baseline and the 12th, 24th month after entering the cohort
  Parameters from echocardiogram will be collected including posterior wall thickness in millimeter, septal thickness in millimeter, Left Ventricle Length in millimeter, Left Atrium length in millimeter, Left Ventricle Mass in gram, left ventricular diastolic volume in milliliter, left ventricular systolic volume in milliliter, left ventricular ejection fraction in percent, ejection volume in milliliter and E/A ratio.
Change from baseline in levels of Mini-Mental State Examination(MMSE) in 2 years | Baseline and the 12th, 24th month after entering the cohort
  The Mini-Mental State Examination (MMSE) is a widely used tool for assessing cognitive function. It is commonly employed in clinical and research settings to screen for cognitive impairment, monitor cognitive changes over time, and assess the severity of cognitive dysfunction.The MMSE has a minimum score of 0 and a maximum score of 30. Higher scores indicate better cognitive function, while lower scores suggest greater cognitive impairment.
  General guidelines for interpreting MMSE scores are:
  * 24-30: No cognitive impairment
  * 18-23: Mild cognitive impairment
  * 0-17: Severe cognitive impairment
Change from baseline in levels of Montreal Cognitive Assessment (MoCA) in 2 years | Baseline and the 12th, 24th month after entering the cohort
  The MoCA is a screening tool for detecting mild cognitive impairment (MCI) and early dementia.The MoCA has a maximum score of 30. A score of 26 or higher generally indicates normal cognitive function.Scores below 26 suggest varying degrees of cognitive impairment, though age, education, and cultural differences can affect interpretation. Higher scores reflect better cognitive performance. Lower scores indicate greater cognitive impairment.
Change from baseline in levels of Auditory Verbal Learning Test-H (AVLT-H) in 2 years | Baseline and the 12th, 24th month after entering the cohort
  The AVLT-H is used to evaluate verbal memory, learning, and recall. It is a variant of the traditional AVLT adapted for specific populations. It assesses immediate recall, delayed recall, and recognition memory through a list-learning paradigm.The total score depends on the number of correct responses during the recall and recognition phases. Higher scores indicate better memory performance and learning ability.
Change from baseline in levels of Trail Making Test-B (TMT-B) in 2 years | Baseline and the 12th, 24th month after entering the cohort
  TMT-B measures executive function, specifically cognitive flexibility, attention, and task-switching ability.The score is the time taken (in seconds) to complete the task. Errors must be corrected, which can increase the time. Lower scores (shorter completion time) indicate better executive function. Higher scores (longer completion time) suggest poorer cognitive flexibility or attention.
Baseline levels of total and phosphorylated Tau | Baseline
  Tau is the marker of neuronal injury and tauopathy. Lower levels are generally not diagnostic but may indicate absence of disease.Total Tau (t-Tau): Reflects overall neuronal injury. Phosphorylated Tau (p-Tau): Specifically associated with Alzheimer's disease pathology.
Baseline plasma levels of Neurofilament Light Chain (NfL) | Baseline
  Non-specific marker of axonal damage, elevated in numerous neurological diseases, including multiple sclerosis (MS), amyotrophic lateral sclerosis (ALS), Alzheimer's, and traumatic brain injury.
Baseline plasma levels of Glial Fibrillary Acidic Protein (GFAP) | Baseline
  Marker of reactive astrocytosis, a process where astrocytes become activated in response to brain injury or disease. Elevated in conditions with neuroinflammation, such as MS, traumatic brain injury, and Alzheimer's.

CONTACTS AND LOCATIONS:
Locations (1):
- Ruijin Hospital - Shanghai Jiaotong University School of Medicine, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No
Due to concerns regarding patient privacy and hospital policy restrictions, there are currently no plans to make individual participant data (IPD) publicly available.